CLINICAL TRIAL: NCT01855256
Title: Treatment of Hyperhidrosis With Oxybutynin: a Randomized Controlled Double Blind Against Placebo
Brief Title: Treatment of Hyperhidrosis With Oxybutynin
Acronym: H²O
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RB 12.035 H²O
Record Dates: First submitted 2013-05-13; First posted 2013-05-16 (Estimated); Last update posted 2025-12-03 (Actual); Status verified 2014-07

CONDITIONS: Hyperhidrosis
Keywords: hyperhidrosis; oxybutynin
MeSH Terms: conditions — Hyperhidrosis | interventions — oxybutynin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- oxybutynin (Experimental): Oxybutynin was done at 2.5 mg/day from day 1 to day 4, then at 5 mg/day from day 5 to day 7 and at 7.5 mg/day from day 8 to the end of the 6 weeks.
  Interventions: Drug: Oxybutynin
- Placebo (Placebo Comparator): Placebo was done at 2.5 mg/day from day 1 to day 4, then at 5 mg/day from day 5 to day 7 and at 7.5 mg/day from day 8 to the end of the 6 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxybutynin — Oxybutynin is started at a dose of 2.5 mg / day and increased gradually until an effective dose without exceed 7.5 mg / day up to 6 weeks.
  Arms: oxybutynin
Drug: Placebo — Placebo is started at a dose of 2.5 mg / day and increased gradually until an effective dose without exceed 7.5 mg / day up to 6 weeks.
  Arms: Placebo

SUMMARY:
Evaluation of the effectiveness of oxybutynin in hyperhidrosis

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years
* Patient affiliated to social security or beneficiary of such a regime
* Patient able to consent
* Patient with hyperhidrosis, generalized or localized (palmar, plantar, axillary) and whose score HDSS (Hyperidrosis Disease Severity Scale) is greater than two.

Exclusion Criteria:

* Age less than 18 years
* Patient who can't be followed
* Patient participating in another clinical trial
* Pregnant
* Woman breastfeeding
* Hypersensitivity to oxybutynin or any of the excipients
* Risk of urinary retention related disorders uretroprostatiques
* Intestinal obstruction
* Toxic megacolon
* Intestinal atony
* Severe Ulcerative Colitis
* Myasthenia
* Closure glaucoma the anterior chamber angle or slightly deep

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2013-06; Primary Completion 2014-02 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Evaluation of the effectiveness of oxybutynin in hyperhidrosis | 6 weeks
  Two scales are used for this evaluation (Hyperhydrosis Disease Severity Scale and Dermatology Life Quality Index )

SECONDARY OUTCOMES:
Safety evaluation of treatment in this indication | 6 weeks
  Number of Participants with Adverse Events will be followed.

CONTACTS AND LOCATIONS:
Overall Officials: Martine SCHOLLHAMMER, MD, Principal Investigator — ADBO
Locations (4):
- France (4):
  - CHG de Morlaix, Morlaix, France
  - Hospital, Brest, Brest
  - CHG Landerneau, Landerneau
  - Dermatologist'S Office, Quimper

REFERENCES:
- [Result] Schollhammer M, Brenaut E, Menard-Andivot N, Pillette-Delarue M, Zagnoli A, Chassain-Le Lay M, Sassolas B, Jouan N, Le Ru Y, Abasq-Thomas C, Greco M, Penven K, Roguedas-Contios AM, Dupre-Goetghebeur D, Gouedard C, Misery L, Le Gal G. Oxybutynin as a treatment for generalized hyperhidrosis: a randomized, placebo-controlled trial. Br J Dermatol. 2015 Nov;173(5):1163-8. doi: 10.1111/bjd.13973. Epub 2015 Oct 14. PMID 26114588